CLINICAL TRIAL: NCT06724601
Title: Lung Volume Changes in Stable Preterm Infants Positioned in Car Seats - A Prospective Observational Study
Brief Title: Lung Volume Changes in Stable Preterm Infants Positioned in Car Seats
Acronym: CarSeat
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: CarSeat
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Premature Birth; Electrical Impedance Tomography (EIT); Lung Volume; Car Seat Transition for At-risk Infants
Keywords: electrical impedance tomography; premature birth; car seat
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Preterm infants < 37 weeks gestation at birth or birthweight <2.5 kg (within 48 hours of discharge): Preterm infants with gestational age up to 36 6/7 weeks at birth and/or birthweight < 2.5 kg will be included. They must fulfill all criteria for discharge from the Neonatal Intensive Care Unit and be discharged home within 48 hours at the time of measurement.
  Interventions: Device: Electrical Impedance Tomography

INTERVENTIONS:
Device: Electrical Impedance Tomography — Electrical Impedance Tomography data and the physiological and clinical parameters will be recorded continuously in three different positions (supine 1, car seat, supine 2) to assess alterations in lung volume and cardiorespiratory events.

SUMMARY:
Premature infants (infants born <37 weeks' gestational age) are discharged from the hospital and transported home in car seats designed for term babies. The safe transport of these premature infants is an important concern. Sub-optimal positioning in car seats can lead to breathing problems in premature infants. With the help of electrical impedance tomography, the investigators want to assess the changes in lung volume during the transition from a supine to a semi-upright position in the car seat.

DETAILED DESCRIPTION:
Hypothesis The investigators hypothesise that there is a decrease in the end-expiratory lung volume (EELV) of preterm infants transferred from supine to car seat position. They expect that the curved, semi-upright built of a standard car seat negatively impacts lung aeration and ventilation of preterm infants, which may result in cardiorespiratory events. They also hypothesise that EELV will normalise following the repositioning of the infant back to the supine position.

Primary objective The primary objective of this study is to assess lung volume changes during the transition from a supine to a semi-upright position in a car seat in preterm infants.

Study procedures As soon as all inclusion criteria are met, the study intervention is initiated. For the baseline measurement, the child is placed in supine position on a flat surface. The EIT belt is attached at nipple level around the infant's thorax during the last nursing care before the start of the intervention. Continuous measurement is conducted for 30 minutes.

Subsequently, the child, with the EIT belt securely in place, is repositioned from a supine to a semi-upright position in a car seat, where another 30-minute measurement is taken. A third measurement will be conducted after the infant is returned to the standard supine position in his/her cot. Manipulations during the measurement periods will be kept to a minimum to avoid disruptions or artefacts in the data recordings. EIT data will be obtained for a total of 90 minutes (plus a maximum of 10 minutes for repositioning).

Subgroup analyses will be performed for the primary outcome:

* Preterm infants ≥ 32 versus < 32 weeks at birth
* Infants with a weight ≥ 2 kg versus < 2 kg at the time of the study
* Car seat positioning: nursing staff versus parents

ELIGIBILITY:
Inclusion Criteria:

* Gestational age up to 36 6/7 weeks at birth and/or birthweight < 2.5 kg
* Preterm born infants fulfilling all criteria for discharge from the NICU
* Discharge home planned within 48 hours
* Written informed consent by one or both parents or legal guardians as documented by signature.

Exclusion Criteria:

* Severe malformation adversely affecting lung aeration or malformations limiting life expectancy.
* Inability of the parents to understand the study procedures due to cognitive or linguistic reasons.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will take place at the Department of Neonatology of the University Hospital Zurich. Preterm infants ready for discharge will be screened for eligibility and parents will be approached by the treating physician or a clinician-researcher who is authorized to access the patient's clinical data.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2025-01-03 (Actual); Primary Completion 2025-08-22 (Actual); Study Completion 2025-08-22 (Actual)

PRIMARY OUTCOMES:
Global end-expiratory lung impedance | Continuous measurement is conducted for 30 minutes in a supine position, 30 minutes in a semi-upright car seat position and an additional 30 minutes in a supine position. Total measurement of 90 minutes.
  Changes in global end-expiratory lung impedance (EELZ) between a baseline measurement in supine position, measurement in a semi-upright car seat position, and a follow-up measurement back in a supine position, as a measure of lung aeration and a proxy for end-expiratory lung volume (∆EELZ = EELZCarSeat - EELZBaseline).

SECONDARY OUTCOMES:
Heart rate | Continuous measurement is conducted for 30 minutes in a supine position, 30 minutes in a semi-upright car seat position and an additional 30 minutes in a supine position. Total measurement of 90 minutes.
  Changes of heart rate between baseline, a semi-upright car seat position, and a follow-up supine position.
Number of bradycardia | Continuous measurement is conducted for 30 minutes in a supine position, 30 minutes in a semi-upright car seat position and an additional 30 minutes in a supine position. Total measurement of 90 minutes.
  Changes in the number of bradycardia (heart rate < 80 bpm) between a baseline measurement in supine position, measurement in a semi-upright car seat position, and a follow-up measurement back in a supine position.
Respiratory rate | Continuous measurement is conducted for 30 minutes in a supine position, 30 minutes in a semi-upright car seat position and an additional 30 minutes in a supine position. Total measurement of 90 minutes.
  Changes in respiratory rate between baseline, a semi-upright car seat position, and a follow-up supine position based on EIT data.
Oxygen Saturation | Continuous measurement is conducted for 30 minutes in a supine position, 30 minutes in a semi-upright car seat position and an additional 30 minutes in a supine position. Total measurement of 90 minutes.
  Changes in oxygen saturation between baseline, a semi-upright car seat position, and a follow-up supine position.
Number of desaturations | Continuous measurement is conducted for 30 minutes in a supine position, 30 minutes in a semi-upright car seat position and an additional 30 minutes in a supine position. Total measurement of 90 minutes.
  Changes in the number of desaturations (SpO2 < 80%) between a baseline measurement in supine position, measurement in a semi-upright car seat position, and a follow-up measurement back in a supine position.
Regional end-expiratory lung impedance | Continuous measurement is conducted for 30 minutes in a supine position, 30 minutes in a semi-upright car seat position and an additional 30 minutes in a supine position. Total measurement of 90 minutes.
  Changes in regional end-expiratory lung impedance between baseline, a semi-upright car seat position, and a follow-up supine position.
Tidal Volume | Continuous measurement is conducted for 30 minutes in a supine position, 30 minutes in a semi-upright car seat position and an additional 30 minutes in a supine position. Total measurement of 90 minutes.
  Changes in tidal volume using EIT between baseline, a semi-upright car seat position, and a follow-up supine position.
Respiratory minute volume | Continuous measurement is conducted for 30 minutes in a supine position, 30 minutes in a semi-upright car seat position and an additional 30 minutes in a supine position. Total measurement of 90 minutes.
  Changes in respiratory minute volume using EIT between baseline, a semi-upright car seat position, and a follow-up supine position.
Regional tidal volume distribution | Continuous measurement is conducted for 30 minutes in a supine position, 30 minutes in a semi-upright car seat position and an additional 30 minutes in a supine position. Total measurement of 90 minutes.
  Changes in regional tidal distribution using EIT between baseline, a semi-upright car seat position, and a follow-up supine position.
Silent spaces, depenent | Continuous measurement is conducted for 30 minutes in a supine position, 30 minutes in a semi-upright car seat position and an additional 30 minutes in a supine position. Total measurement of 90 minutes.
  Changes in dependent silent spaces using EIT between baseline, a semi-upright car seat position, and a follow-up supine position.
Silent spaces, nondependent | Continuous measurement is conducted for 30 minutes in a supine position, 30 minutes in a semi-upright car seat position and an additional 30 minutes in a supine position. Total measurement of 90 minutes.
  Changes in nondependent silent spaces using EIT between baseline, a semi-upright car seat position, and a follow-up supine position.
Center of ventilation, ventral to dorsal | Continuous measurement is conducted for 30 minutes in a supine position, 30 minutes in a semi-upright car seat position and an additional 30 minutes in a supine position. Total measurement of 90 minutes.
  Changes in center of ventilation (ventral to dorsal) using EIT between baseline, a semi-upright car seat position, and a follow-up supine position.
Center of ventilation, left to right | Continuous measurement is conducted for 30 minutes in a supine position, 30 minutes in a semi-upright car seat position and an additional 30 minutes in a supine position. Total measurement of 90 minutes.
  Changes in center of ventilation (left to right) using EIT between baseline, a semi-upright car seat position, and a follow-up supine position.
Global inhomogeneity index | Continuous measurement is conducted for 30 minutes in a supine position, 30 minutes in a semi-upright car seat position and an additional 30 minutes in a supine position. Total measurement of 90 minutes.
  Changes in global inhomogeneity index using EIT between baseline, a semi-upright car seat position, and a follow-up supine position.
Coefficient of variation | Continuous measurement is conducted for 30 minutes in a supine position, 30 minutes in a semi-upright car seat position and an additional 30 minutes in a supine position. Total measurement of 90 minutes.
  Changes in coefficient of variation using EIT between baseline, a semi-upright car seat position, and a follow-up supine position.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Bassler, Prof., Study Chair — Newborn Research, Department of Neonatology, University Hospital and University of Zurich, Zurich, Switzerland
Locations (1):
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No